CLINICAL TRIAL: NCT04502875
Title: A Randomized, Double-blind Controlled Trial to Evaluate the Efficacy of Intracavernosal Infusion of Platelet Rich Plasma Against Platelet Poor Plasma in the Treatment of Vasculogenic Erectile Dysfunction.
Brief Title: Clinical Trial to Evaluate the Efficacy of Intracavernosal Infusion of PRP vs PPP for the Erectile Dysfunction.
Acronym: PRePED
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Juan Ignacio Martinez Salamanca, Principal Investigator, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRePED
Record Dates: First submitted 2020-07-16; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Erectile Dysfunction
Keywords: Platelet Rich Plasma; Platelet Poor Plasma
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind clinical trial to evaluate efficacy, feasibility and safety with two groups in a 1:1 ratio; where the control group corresponds to patients who will receive PPP and an experimental group where patients will receive PRP, both collected by apheresis.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Intracavernosal infusion of Platelet Rich Plasma
  Interventions: Drug: PRP
- Control Arm (Active Comparator): Intracavernosal infusion of Platelet Poor Plasma
  Interventions: Drug: PPP

INTERVENTIONS:
Drug: PRP — Platelet Rich Plasma (PRP) is an autologous blood component derivate from the own patient blood, with a high concentration in platelets. The liquid fraction obtained after the soft centrifugation of Whole Blood (WB) collected with anticoagulant, in a way that most of the red cells and leukocytes are sedimented and removed, but most of the platelets are kept in the supernatant plasma. The platelet concentration in PRP is not well defined.
  Arms: Treatment Arm
Drug: PPP — PPP is the liquid fraction obtained after the hard centrifugation of WB collected with any anticoagulant. PPP does not contain cells. (Hematocrit lower than 1% and leukocytes below 1 x 109/L) x but contains WB proteins (including clotting factors), ions, microelements and water. PPP can be also being collected using an apheresis technique.
  Arms: Control Arm

SUMMARY:
Randomized, double-blind clinical trial to evaluate efficacy, feasibility and safety with two groups in a 1:1 ratio; where the control group corresponds to patients who will receive Platelet Poor plasma and an experimental group where patients will receive Platelet Rich Plasma, both collected by apheresis.

DETAILED DESCRIPTION:
Patients treated in the urology department of the Hospital Universitario Puerta de Hierro Majadahonda, are eligible and will be offered the participation in this clinical trial.

The target populations are patients who presented erectile dysfunction for at least 6 months with an IIEF-EF between 5 and 16 points. They will be pre-screened for eligibility.

The patient must complete the informed consent form (ICF) process and sign and date the informed consent form prior to participation in this study, including completion of any non-standard-of- care procedures required for this clinical Investigation.

If the patient meets the inclusion criteria and additionally meet with the apheresis procedures, the patient wil be included in the study.

The study include two phases. In the first phase, the patient will be randomized to PPP or PPP. In the second phase, according with the score IIEF-EF (responder or non responder), the patient will receive PRP.

With the responders patients, an open phase with PDE5-Is is initiated. The patient will use phosphodiesterase 5 inhibitors (PDE5-Is) at maximum tolerated doses according with the Summary Product of characteristics.

With the no responders patients, there will be two options:

If the non-responder patient was in treatment with PRP during the firs phase, the patient will continue with the procedures of visits 11a and 12a.

If the non-responder patient was in treatment with PPP, the patient will start the second phase of treatment with PRP and will continue with the procedures of this treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Signed an ethics committee-reviewed and approved informed consent form.
* Subjects must meet all inclusion criteria to be eligible for study enrollment.
* Men between 40 and 75 years old, with a relationship of more than 6 months of duration.
* Erectile dysfunction for at least 6 months with an IIEF-EF (while using the higher tolerated dose of PDE5-Is) between 5 and 16 points, inclusive.
* Erectile dysfunction of vascular origin. In case of clinical doubt or incongruence, a Nocturnal Penile Tumescence and Rigidity Test (NPTR) will be performed. In this case, criteria inclusion is having no event in the night with a penile rigidity (tip) of ≥70% during ≥5min.
* Subjects agree to attempt vaginal intercourse at least 4 times every month after the end of the treatment and agree to document the outcome using the Sexual Encounter Profile (SEP) and the Erection Hardness Score (EHS).
* Commitment not to use other treatment for ED during the study (herbal, topical, intraurethral, intracavernosal, etc.).
* Commitment to completing the rest of the questionnaires and other measurement instruments during the study phase.
* Willingness and ability to comply with study procedures, other measurements instruments and visit schedules and able to follow oral and written instructions.

Exclusion Criteria:

* Documented psychogenic erectile dysfunction (with NPTR test: at least one event in the night with a penile rigidity (tip) of ≥70% during ≥5min).
* Erectile dysfunction of neurogenic origin (radical prostatectomy, pelvic surgery, spinal cord injury, multiple sclerosis, diabetes mellitus is not included unless documented diabetic neuropathy).
* Some other current sexual dysfunction (premature ejaculation, etc.).
* Prior implant of penile prosthesis or other penile surgeries different to circumcision, frenuloplasty or condyloma removal.
* Previous history of penile fracture, Peyronie's disease or priapism.
* History of radical prostatic or bladder surgery (radical cystectomy or prostatectomy).
* Previous radiation to pelvis.
* History of symptomatic hypogonadism (testosterone level <346ng/dl) not treated. If treated hypogonadism, testosterone levels non-stable for at least 3 months.
* Major hematologic, renal, or hepatic abnormalities.
* Severe decompensated cardiac and vascular insufficiency, or critical coronary heart disease.
* Poorly controlled hypertension or diabetes mellitus (HbA1c >12%).
* Recent (within previous six months of the inclusion) stroke or myocardial infarction.
* Active peptic ulcer disease.
* Neoplasm of any origin in active treatment or active progression.
* History of psychiatric pathology (depressive syndrome, schizophrenia, bipolar disorder).
* History of alcohol abuse (More than 7 alcohol drink units a week or more than 3 per occasion) or drug abuse (any drug consumption different to alcohol or tobacco, used more than three times per month).
* Treatment with oral anticoagulants (dicoumarin or by-products) or antiandrogens.
* Active treatment as nitric oxide (NO) donor drugs.
* Prior positive serology to HBsAg, HCV (by genomic test), HIV-1/2, syphilis.
* Thrombopenia less than 100 x 109 / L.
* Anemia (Hemoglobin <13 g/dl).
* Poor venous access or any other circumstance that preclude an apheresis procedure.
* Lack of sexual practices in recent months (less than 4 attempts in the last three months).
* Lack of commitment on the part of the patient to attend the tests requested.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference of increments between PRP and PPP treatment assessed by IIEF scale | 28 weeks
  Difference of increments between both treatment groups assesed by International Index Erectile Function (IIEF) scale (referred to the investigator's study as mean PRP V9(PT)IIEF-EF - V3IIEF-EF vs mean PPP V9(PT)IIEF-EF - V3IIEF-EF) after 4 weeks of the end of the treatment.

SECONDARY OUTCOMES:
Incidence of adverse events related with the use of PRP/PPP | 28 weeks
  Incidence of infusion related Adverse Events (AEs) and cumulative of incidence of Serious Adverse Events (SAEs) during the clinical trial.
Synergic efficcacy of PRP and PDE5 inhibitors | 28 weeks
  Assessment of the synergic efficacy of PRP treatment on the therapeutic response to oral administration of PDE5 inhibitors by the IIEF.
Concentration of cytokines and growth factors in the PRP and PPP | 28 weeks
  Concentration of cytokines and growth factors concentration in the PRP and PPP of each patient and their relationship with the clinical response to PRP assessed by IIEF.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Martinez-Salamanca, Md, PhD, Principal Investigator — Urologist
Locations (1):
- Puerta de Hierro University Hospital, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No